CLINICAL TRIAL: NCT00213889
Title: TWIST Human Gene and Cleft Lips and Palates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2602
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Cleft Lip
Keywords: Facial clefting; twist; craniofacial development genes; Human cleft lip and palate; cleft lip and palate
MeSH Terms: conditions — Cleft Lip; Acrocephalosyndactylia

INTERVENTIONS:
Other: None: molecular genetics diagnosis procedure only — None: molecular genetics diagnosis procedure only

SUMMARY:
This study uses a sequence analysis for TWIST and other craniofacial development genes, among patients presenting with facial clefting.

ELIGIBILITY:
Inclusion Criteria:

Patients aged from 1 month to 18 years:

* Parents agree to enrollment or patients, themselves, agree to enrollment when able to do so
* Healthcare insurance holders
* Display facial clefting

Grown patients over 18 years of age:

* Agree to enrollment
* Display facial clefting
* Healthcare insurance holders

Exclusion Criteria:

* Patients declining enrollment
* Patients without healthcare insurance

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
to show, among patients displaying facial clefting, the TWIST mutations and the mutation in genes involved with TWIST in craniofacial development | Not relevant

SECONDARY OUTCOMES:
to show, among patients displaying facial clefting and mutations in such genes, possible mutations in the same genes | Not relevant

CONTACTS AND LOCATIONS:
Overall Officials: Pascal TSCHILL, MD, Principal Investigator — Laboratoire de Génétique Molécules des Eucaryotes (LGME)
Locations (4):
- France (4):
  - Centre d'Investigations Cliniques, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre de Soins , d'Enseignement et de Recherche Dentaire (CESRD), Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Chirurgie Infantile, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Consultation de la Face, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg